CLINICAL TRIAL: NCT02651480
Title: A Nutritional Intervention in Police Officers
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor put plans on hold
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: Metropolitan Police Department of Washington, D.C. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PCRM MPD
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Overweight; Blood Pressure; Diabetes Mellitus, Type 2
Keywords: Diet, Vegetarian; Diet, Fat-Restricted; Quality of Life; Glycemic Index
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 2 | interventions — Diet, Plant-Based; Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vegan Group (Experimental): Participants in the intervention group will follow a low-fat, plant-based diet for 14 weeks, and will attend nutrition classes in the form of a weekly support group.
  Interventions: Dietary Supplement: Plant-based diet
- Control Group (Active Comparator): The control group will follow an unrestricted diet with no instruction.
  Interventions: Dietary Supplement: Control Group

INTERVENTIONS:
Dietary Supplement: Plant-based diet — Weekly instructions will be given to the participants in the intervention group about following vegan diet.
  Other Names: Vegan Group
  Arms: Vegan Group
Dietary Supplement: Control Group — Unrestricted diet with no instruction.
  Other Names: Control
  Arms: Control Group

SUMMARY:
The proposed study seeks to test the effect of a plant-based dietary intervention on cardiovascular risk factors in police officers.

DETAILED DESCRIPTION:
This study tests the hypotheses that a low-fat, plant-based (vegan) diet improves body weight, plasma lipid concentrations, blood pressure, and, in individuals with type 2 diabetes, glycemic control, that a low-fat, plant-based diet improves health-related quality of life as measured by the Medical Outcomes Study Short Form 36-Item Health Survey (SF-36), and that a low-fat, plant-based diet improves mood, as measured by the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years
2. Body mass index ≥ 25 kg/m2 and/or a diagnosis of type 2 diabetes mellitus, as defined by a fasting plasma glucose concentration ≥ 126 mg/dl on two occasions or a prior physician's diagnosis of type 2 diabetes
3. Currently an employee of the Metropolitan Police Department of the District of Columbia
4. Ability and willingness to participate in all components of the study
5. A willingness to be randomly assigned to either study group

Exclusion Criteria:

1. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
2. Use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
3. Pregnancy
4. Unstable medical or psychiatric illness
5. Likely to be disruptive in group sessions (as determined by research staff)
6. Already following a low-fat, vegan diet
7. Lack of English fluency
8. Inability or unwillingness to participate in all components of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Changes in body weight from Baseline at 14 weeks
  body weight will be measured to the nearest 0.1 kg, using a digital scale.
Plasma lipid concentrations | Changes in plasma lipid concentrations from Baseline at 14 weeks
  will be measured using the Olympus Cholesterol Reagent on Olympus Chemistry Analyzers to assess changes in plasma lipid concentrations.
Blood pressure | Changes in blood pressure from Baseline at 14 weeks
  Blood pressure will be measured at each assessment

SECONDARY OUTCOMES:
Quality of Life and Mood | Change in quality of life from Baseline at 4 months
  Measured by a Modified Health Assessment Questionnaire (MHAQ). The questionnaire measures the difficulty level of performing 8 different activities. A score of 0 = the activity can be performed without difficulty. A score of 3 = the activity cannot be performed. The MHAQ is calculated as the average of these scores.

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Barnard, M.D., Principal Investigator — President
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No